CLINICAL TRIAL: NCT05913492
Title: Difficult Airway Simulation-based Training in Anaesthesiologists: Efficacy and Skills Retention Within Six Months After Training
Brief Title: Difficult Airway Simulation-based Training
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Associated professor at the Department of OF SURGERY, ANESTHESIOLOGY AND INTENSIVE THERAPY OF POSTGRADUATE EDUCATION, Bogomolets National Medical University
Other Study IDs: 4012
Record Dates: First submitted 2023-05-15; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Intubation; Difficult or Failed; Educational Problems; Critical Illness
Keywords: difficult airways; simulation training
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Each volunteer went through two simulation scenarios of difficult airway management on the first time
- Group 2: Each volunteer went through two simulation scenarios of difficult airway management after training in difficult airway management according to DAS guidelines, using the same equipment as during the simulation
  Interventions: Behavioral: Simulation training
- Group 3: Each volunteer went through two simulation scenarios of difficult airway management after 6 month
  Interventions: Behavioral: Simulation training

INTERVENTIONS:
Behavioral: Simulation training — Each volunteer went through two simulation scenarios of difficult airway management: 1) "cannot intubate, can ventilate" (CI), 2) "cannot intubate, cannot ventilate" (CICV) with the assistance of the training centre operator. Following the first simulation round, volunteers were trained on the same day in difficult airway management according to DAS guidelines, using the same equipment as during the simulation. The participants repeated the simulation scenarios immediately after the training and six months later.
  Groups: Group 2; Group 3

SUMMARY:
Difficult airways remain a significant problem in anaesthesia, intensive care and emergency medicine. Simulation-based training gives better outcomes compared to non-simulation and non-intervention education. However, it remains unclear how long the acquired skills are retained and how often simulation training should repeat. The study aimed to investigate the efficacy and skills retention in training for difficult airway management in anaesthesiologists. After ethical committee approval, we conducted a prospective control study at the postgraduate Department of Surgery, Anaesthesiology and Intensive Therapy (Bogomolets National Medical University) from July to December 2022. Anaesthesiologists who applied for the continuous medical education course "Difficult airways management" were involved in the study. The simulation room included a mannequin Laerdal SimMom Advanced Patient Simulator, vital monitor, anaesthesia station LEON and airway devices. Each volunteer went through two simulation scenarios of difficult airway management: 1) "cannot intubate, can ventilate" (CI), 2) "cannot intubate, cannot ventilate" (CICV) with the assistance of the training centre operator. The primary endpoints included: more than three laryngoscopy attempts; supraglottic airway attempt missing; call for help skip; failure to initiate a surgical airway (for the CICV scenario). Secondary endpoints included: time to call for help; mean duration of desaturation; use of bougie; use of video laryngoscope (Airtraq); mean number of intubation attempts; improper usage of equipment of equipment, time to initiation of surgical airway preparation; time to initiation of surgical airway ventilation.

DETAILED DESCRIPTION:
After ethical committee approval, we conducted a prospective control study at the postgraduate Department of Surgery, Anaesthesiology and Intensive Therapy (Bogomolets National Medical University) from July to December 2022. Anaesthesiologists who applied for the continuous medical education course "Difficult airways management" were involved in the study. We obtained consent from them to participate anonymously as volunteers. Before the first training, we interviewed all participants about their experience in working in the speciality, difficult airways management, learning at any simulation training and difficult airways training particularly.

The simulation room included a mannequin Laerdal SimMom Advanced Patient Simulator, vital monitor, anaesthesia station LEON and airway devices. Standard settings included modelling of tongue oedema to grade 4 visualizations on laryngoscopy according to the Cormack and Lehane classification, as well as additional pharyngeal obstruction and stiffness of both lungs for the "cannot ventilate" scenario. A standard set of tools and equipment for ensuring airway patency, ventilation and tracheal intubation included facemasks, oropharyngeal and nasal airways, laryngoscopes, laryngeal masks, and tracheal tubes in a range of sizes. The trolley for difficult airways was available for each station and was equipped with additional laryngoscope blades of various sizes, a video laryngoscope, laryngeal masks of various sizes (Igel), introducers for tracheal tubes (stylets and bougies), Airtraq, a cricotomy kit.

Monitoring provided SpO2, EtCO2, ECG and non-invasive blood pressure measurement. When the oxygen delivery was interrupted for 20 seconds or more, the SpO2 gradually decreased by 3% every 5 seconds and reached 90% after 20 seconds. A value of SpO2 < 90% was considered desaturation. Effective ventilation was defined after at least two effective breaths evidenced by an EtCO2 curve on the monitor.

Each volunteer went through two simulation scenarios of difficult airway management: 1) "cannot intubate, can ventilate" (CI), 2) "cannot intubate, cannot ventilate" (CICV) with the assistance of the training centre operator. Participants were expected to follow an algorithm according to the Difficult Airway Society (DAS) recommendations [4].

During the scenario, we recorded significant deviations from the DAS protocol and other indicators that impacted the quality of the algorithm execution. The primary endpoints included significant deviations from the DAS protocol: more than three laryngoscopy attempts; supraglottic airway attempt missing; call for help skip; failure to initiate a surgical airway (for the CICV scenario). Secondary endpoints included: time to call for help; mean duration of desaturation; use of bougie; use of video laryngoscope (Airtraq); mean number of intubation attempts; improper usage of equipment of equipment, time to initiation of surgical airway preparation; time to initiation of surgical airway ventilation Following the first simulation round, volunteers were trained on the same day in difficult airway management according to DAS guidelines, using the same equipment as during the simulation. The participants repeated the simulation scenarios immediately after the training and six months later. The primary and secondary endpoints were compared between three rounds: initial simulation (Group 1), immediately after training (Group 2), and six months after training (Group 3).

Statistical analysis was performed using licensed Microsoft Office Excel and web source www.socscistatistics.com. We used Student's, Kruskal-Wallis and Fisher's exact tests. The difference was considered significant at α < 5% (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

Adult anesthesiologists volunteers

Exclusion Criteria:

Refusion to participate, age more than 70 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult anesthesiologists volunteers
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Significant deviations from the DAS protocol | 2 hours
  more than three laryngoscopy attempts

SECONDARY OUTCOMES:
Other deviations from DAS protocol | 2 hours
  use of bougie

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bielka K, Kuchyn I, Fomina H, Khomenko O, Kyselova I, Frank M. Difficult airway simulation-based training for anaesthesiologists: efficacy and skills retention within six months. BMC Anesthesiol. 2024 Jan 31;24(1):44. doi: 10.1186/s12871-024-02423-x. PMID 38297196